CLINICAL TRIAL: NCT05249257
Title: A Phase 2, Multicenter, Observational Study to Assess the Durability and Safety of Collagenase Clostridium Histolyticum Injected With GRID Technique in Buttocks or Thigh Cellulite With Laxity in Adult Females
Brief Title: Durability and Safety of CCH With Two Different Injection Techniques in Cellulite With Laxity
Status: Completed | Type: Observational
Sponsor: Endo Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: EN3835-225
Record Dates: First submitted 2022-01-25; First posted 2022-02-21 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2023-01

CONDITIONS: Cellulite; Laxity; Skin; Edematous Fibrosclerotic Panniculopathy
MeSH Terms: conditions — Cellulite; Cutis Laxa

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- No Treatment - previously treated in parent study: Participants who completed the parent study EN3835-224 (NCT04580303) will be eligible for this study.

SUMMARY:
All participants who completed the EN3835-224 study will be invited to participate in this observational study to evaluate long term durability of response and safety.

ELIGIBILITY:
Inclusion Criteria:

1. Have participated in and completed study EN3835-224 (parent study).
2. Be willing and able to cooperate with the requirements of the study.

Exclusion Criteria:

1. Has received any collagenase treatments (eg, Santyl® Ointment) at any time since
2. Has had any surgery, invasive procedure (eg, liposuction), injectable treatment (eg, KYBELLA®) or any similar treatment in the area treated during the EN3835-224 study since the completion of that study.
3. Has any other conditions that, in the investigator's opinion, might indicate the participant to be unsuitable for the study

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The Safety Population is defined as all participants who meet the inclusion/exclusion criteria at Day 360. All Safety analyses will be based on this population.
  The Full Analysis Set (FAS) is defined as all participants in the Safety Population who have at least 1 I-GAIS assessment. All efficacy analyses will be based on this population.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2022-01-25 (Actual); Primary Completion 2022-09-12 (Actual); Study Completion 2022-09-12 (Actual)

PRIMARY OUTCOMES:
Proportion of 1-level responders (+1 or better score) on the I-GAIS for either buttock or either thigh | Day 360
  Investigator Global Aesthetic Improvement Scale (I-GAIS) is a 7-level scale ranging from "+3" (very much improved) to "-3" (very much worse) to determine the degree of improvement of the treated areas
Proportion of 1-level responders (+1 or better score) on the I-GAIS for either buttock or either thigh | Day 540
  Investigator Global Aesthetic Improvement Scale (I-GAIS) is a 7-level scale ranging from "+3" (very much improved) to "-3" (very much worse) to determine the degree of improvement of the treated areas

SECONDARY OUTCOMES:
I-GAIS ratings | Day 360 and Day 540
  Investigator Global Aesthetic Improvement Scale (I-GAIS) is a 7-level scale ranging from "+3" (very much improved) to a "-3" (very much worse) to determine the degree of improvement of the treated areas.
Proportion of 1-level responders (+1 or better score) on the S-GAIS for either buttock or either thigh | Day 360 and Day 540
  Subject Global Aesthetic Improvement Scale (S-GAIS) is a 7-level scale ranging from "+3" (very much improved) to a "-3" (very much worse).
Change from Day 1 (pre-treatment) of the parent study and each study visit in Subsection D of the Hexsel CSS | Day 360 and Day 540
  Hexsel CSS is a photonumeric scale that looks at 5 key morphologic features of cellulite using a 4-point scale ranging from "0" (low) to "3" (high).

CONTACTS AND LOCATIONS:
Overall Officials: Karen Chajko, Study Director — Endo Pharmaceuticals
Locations (3):
- United States (3):
  - Endo Clinical Trial Site #2, Coral Gables, Florida
  - Endo Clinical Trial Site #3, Metairie, Louisiana
  - Endo Clinical Trial Site #1, New York, New York

IPD SHARING:
Plan to Share IPD: No